CLINICAL TRIAL: NCT04897555
Title: Evaluation of Low Level Light Therapy (LLLT) as a Primary Therapy for Non-Specific Alopecia of the Eyebrow in Women
Brief Title: LLLT for Alopecia of the Eyebrow in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freedom Laser Therapy, Inc. (Industry)
Responsible Party: Sponsor
Organization: Freedom Laser, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRE0219
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LLLT Active Treatment (Experimental): LLLT Therapy will be administered to the treatment site.
  Interventions: Device: LLLT
- No LLLT Comparator (No Intervention): No LLLT Therapy will be administered to the comparator site.

INTERVENTIONS:
Device: LLLT — This is a low-level light (LED) device configured in the shape of a headband, operating at 650 +/-10 nanometers and 940 +/- 10 nanometers, that contains 12 of each wavelength for a total of 24 LEDs.
  Arms: LLLT Active Treatment

SUMMARY:
The purpose of this research is to study the ongoing effectiveness of a light therapy device for human hair growth. This device, called the iRestore Eyebrow Device, is a type of cold, or non-heat producing light therapy system that will emit light on the hair growth cells within and around the hair follicle. When these cells do not function properly, one may experience common problems such as baldness and thinning or brittle hair. The application of a special category of low-level light to be studied in the project may cause an increase in essential nutrients to the damaged hair follicles and skin cells, leading to a reduction in hair loss and in some cases, possibly leading to re-growth.

DETAILED DESCRIPTION:
This study on LLLT aims to define the safety and physiologic effects that occur when the human hair follicle and surrounding tissue structures are exposed to this type of radiation. Thus far, all reports on the efficacy of laser light and LED light in this area, have been, in large part, unsupported by multi-center, randomized, double blind, controlled studies. To properly identify the effects in human subjects, exposure to LLLT is not sufficient. The analysis of the non-radiated and radiated tissues is required to elucidate the tissue response and efficacy of the laser therapy. The theory that is widely accepted is that the mitochondria are the powerhouse of the stem cells that cause hair growth. The LLLT "turns on" the nutrient pump process that energizes the mitochondria, which leads to an increase in ATP and subsequent reversal of hair follicles from the dormant stage of growth called telogen, to the active growth stage called anagen.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects experiencing any type of non-traumatic eyebrow hair loss.
* Apparent good health.

Exclusion Criteria:

* Previous involvement in other eyebrow hair studies.
* Use of any hair growth agent within the last 4 weeks.
* Evidence of any current viral, fungal or bacterial infection.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in number of terminal hairs | 12 weeks
  Pre & Post treatment terminal hair counts

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bodian, MD, Principal Investigator — Bodian Dermatology Group
Locations (2):
- United States (2):
  - NST Consultants, Inc., Mendham, New Jersey
  - Bodian Dermatology, Great Neck, New York